CLINICAL TRIAL: NCT01922986
Title: Real vs Sham rTMS Combined With Conventional Therapy in Acute Stroke
Brief Title: Repetitive Transcranial Magnetic Stimulation Use in Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acute_rTMS
Record Dates: First submitted 2013-07-26; First posted 2013-08-14 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; hemiplegia; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active rTMS with conventional therapy (Experimental): 20 minutes of active rTMS followed by conventional stroke therapy
  Interventions: Device: active rTMS; Behavioral: conventional stroke therapy
- sham rTMS with conventional therapy (Sham Comparator): 20 minutes of sham rTMS stimulation followed by conventional stroke therapy
  Interventions: Device: sham rTMS; Behavioral: conventional stroke therapy

INTERVENTIONS:
Device: active rTMS — 10 minutes of real high-frequency (6-Hz) rTMS priming (total priming pulses = 600) plus 10 minutes of low-rate (1Hz) rTMS (total low-rate pulses = 600).
  Arms: Active rTMS with conventional therapy
Device: sham rTMS — 20 minutes of sham rTMS stimulation
  Arms: sham rTMS with conventional therapy
Behavioral: conventional stroke therapy — conventional stroke therapy consisting of exercises and physical training

SUMMARY:
When a certain area of the brain is injured, like in stroke, several events occur. One side of the body may become weak. This weakness is called hemiparesis and it may create difficulty in performing tasks like writing, eating, and walking. The weakness results from two sources:

1. death of some brain cells in the affected side (hemisphere) of the brain
2. exaggerated inhibitory signals from the unaffected hemisphere acting on surviving neurons in the affected hemisphere.

Investigators cannot change neurons that have died but they may be able to change the exaggerated inhibition that impairs the surviving neurons in the affected hemisphere.The purpose of this study is to try to decrease the exaggerated inhibition coming from the unaffected hemisphere, which suppresses the affected hemisphere, with transcranial magnetic stimulation (TMS). Investigators hypothesize that, from admission to discharge, active rTMS combined with conventional therapy will produce greater functional gains in the paretic hand compared to sham rTMS combined with conventional therapy, as measured by standard tests.

DETAILED DESCRIPTION:
Stroke is the leading cause of long-term disability in the United States and people with stroke deserve our maximum effort to restore in them as much function as possible; yet, mainstream stroke rehabilitation remains mired in traditional treatment approaches that may be suboptimal. However, for the past 5 years we have been endeavoring to advance stroke rehabilitation by including noninvasive brain stimulation. This study will explore whether the safety and functional results from noninvasive brain stimulation in patients with chronic stroke when given by researchers in a laboratory setting can be replicated in acute stroke when given by trained clinicians in the real-world clinical setting.

As background, a phenomenon in stroke is that compensatory overuse of the non-stroke hemisphere can inhibit surviving neurons in the stroke hemisphere. In this way, people with stroke are "doubly disabled" - first, by the stroke itself and, second, by exaggerated interhemispheric inhibition (IHI) arising in the non-stroke hemisphere and acting on surviving neurons in the non-stroke hemisphere. Investigators cannot bring the killed neurons back to life but they can up-regulate the surviving neurons suppressed by IHI. Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive way to do this.

rTMS has not yet entered mainstream clinical use for stroke, likely because it has not been explored in the acute rehabilitation setting with application by clinicians. With prior National Institutes of Health funding, Dr. Carey has considerable experience in using rTMS in the laboratory setting for chronic stroke. He will now take rTMS out of his lab and into the real-world setting of Courage Kenny Rehabilitation Institute (CKRI), the primary referral center for acute stroke rehabilitation in our region, where clinicians will be trained in rTMS. Five daily rTMS treatments (active or sham) will be given to the non-stroke primary motor area (M1). After each treatment, patients will receive their conventional rehabilitation training. This approach is innovative because of the rTMS parameters used and because the application will be given by trained clinicians with oversight by the Principal Investigator, as opposed to laboratory researchers. Expected outcomes are improved hand function with no major adverse effects. Data will serve as a springboard to larger clinical trials.

Specific Aim #1: Determine the safety of 5 treatments of 6-Hz primed low-frequency rTMS combined with conventional therapy in adults with acute stroke.

Adverse effects will be measured through observation for seizures, investigator screening, physician exam, and tests of cognitive function and motor function in the nonparetic hand.

Investigators hypothesize there will be a) no seizures, b) no cognitive decline and c) no motor decline.

Specific Aim #2: Compare the effectiveness of active vs. sham rTMS on functional outcomes in adults with acute stroke.

Adults with acute stroke will be randomized to receive either active rTMS or sham rTMS. Both groups will also receive conventional therapy, consisting of the normal rehabilitation used at this rehabilitation center. Investigators hypothesize that, from admission to discharge, active rTMS will produce greater functional gains in the paretic hand compared to sham rTMS, as measured by standard tests.

ELIGIBILITY:
Inclusion Criteria:

* stroke onset: within past 30 days but rTMS intervention will commence no sooner than 5 days from stroke onset
* stroke location: cortical or subcortical
* stroke type: ischemic
* age: >18 years
* paretic index finger must show either no or impaired flexion/extension motion at the metacarpophalangeal (MP) joint.
* Mini-Mental State Examination greater than or equal to 22
* ability to stand/transfer with no more than moderate assistance

Exclusion Criteria:

* seizure within past two years
* metal in head (dental permitted)
* pregnancy
* psychiatric disorders
* receiving tricyclic antidepressants or neuroleptics
* inability to follow three-step command
* hemineglect
* dependent on ventilator, nasogastric tube, or implanted medical device
* co-morbidities impairing upper extremity function
* anticipated stay at Courage Kenny Rehabilitation Institute shorter than 7 treatment days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Carey, PhD, PT, Principal Investigator — University of Minnesota
Locations (1):
- Courage Kenny Rehabilitation Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS With Conventional Therapy | Sham rTMS With Conventional Therapy
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Four people with acute stroke were enrolled. All four completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS With Conventional Therapy | Sham rTMS With Conventional Therapy | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (19.1) | 52.5 (23.3) | 63.0 (21.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Jebsen Taylor Hand Function Test Scores
Description: This test quantifies the time it takes for the subject to do the following standardized functional tasks with the hand: stack three checkers, turn over cards, turn over empty cans, turn over fluid-filled cans, pick up and place small items like a paper clip, etc into a can, and use a spoon to scoop up a bean and drop the bean into a can. The unit of measure is time and changes that are negative signify reduced time at posttest compared to pretest, which would be an improvement. Total score = sum of times for each subtests
Time Frame: Measured at pretest (day before treatments begin) and posttest (day following last treatment). Thus, 7 days of participation (1 pretest, 5 treatments, 1 posttest).
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Active rTMS With Conventional Therapy | Sham rTMS With Conventional Therapy
Number analyzed (Participants) | 2 | 2
percentage of change from baseline | -23.0 (32.5) | 0 (0)

2. Secondary Outcome: Change in Finger Tracking Test
Description: This test involves placing a device on the hand that shows the changing angle of the finger joint on a computer screen as the joint is moved. The computer screen also shows a target line, such as a sine wave. At the start of the test, the computer screen cursor moves horizontally across the target and the subject moves the finger joint into extension or flexion to adjust the vertical position of the cursor to that it traces the target line as accurately as possible. The performance is quantified by calculating the root-mean-square error between the target line and the response line. This is converted into an Accuracy Index, which has a maximum value of 100% (perfect score). Negative values can occur and reach a value of -100%, signifying very poor performance. Typical scores for healthy range from 50-80%. Typical values in stroke range from -100 to +40%. Changes that are positive signify increased tracking accuracy at posttest compared to pretest, which would be an improvement.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS With Conventional Therapy | Sham rTMS With Conventional Therapy
Number analyzed (Participants) | 2 | 2
units on a scale | 24.5 (25.2) | -13.8 (41.8)

3. Secondary Outcome: Change in Motricity Index
Description: Measures strength in finger pinch, elbow flexion and arm abduction. 0 No pinch movement. 11 Slight movement of finger or thumb. 19 Able to grip the cube, but not hold it against gravity. 22 Able to grip and hold the cube against gravity, but not against a weak pull by examiner.
  The weighted score based on the ordinal 6 point scale 26 Able to grip and hold the cube against a weak pull, but weaker than the other side.
  33 Normal pinch grip.
  For shoulder and elbow scoring is:
  0 No movement. 9 Palpable contraction in muscle, but no movement. 14 Visible movement, but not full range and not against gravity. 19 Full range of movement against gravity but not against resistance. 25 Full movement against resistance, but weaker than the other side. 33 Normal power. Maximum total score is 99, minimum is 0. Changes that are positive signify improved strength at postte
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS With Conventional Therapy | Sham rTMS With Conventional Therapy
Number analyzed (Participants) | 2 | 2
units on a scale | 4 (5.7) | 11 (0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Active rTMS With Conventional Therapy | Sham rTMS With Conventional Therapy
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Enrollment of subjects was insufficient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No